CLINICAL TRIAL: NCT03881943
Title: A Randomized, Single Center Trial to Assess the Endothelial Function With Ticagrelor Monotherapy Compared to Aspirin Monotherapy in Patients With History of Acute Coronary Syndrome
Brief Title: Ticagrelor Monotherapy Compared to Aspirin Monotherapy in Patients With History of ACS
Acronym: FMD_ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tse Hung Fat, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMD_1.3
Record Dates: First submitted 2019-03-05; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Aspirin; Tablets; Diltiazem

STUDY DESIGN:
Intervention Model Description: Ticagrelor or Aspirin
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor 60mg BD for 3 months
  Interventions: Drug: Ticagrelor 60 mg
- Aspirin (Active Comparator): Aspirin 100mg daily for 3 months
  Interventions: Drug: Aspirin 100 MG Oral Tablet, Enteric Coated

INTERVENTIONS:
Drug: Ticagrelor 60 mg — Potent antiplatelet agent, 60mg twice daily for 3 months
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Aspirin 100 MG Oral Tablet, Enteric Coated — antiplatelet agent, 100mg once daily for 3 months
  Other Names: Cartia
  Arms: Aspirin

SUMMARY:
Antiplatelet agents are cornerstones for management of ischemic heart disease. For patients suffering from acute coronary syndrome (heart attack), treatment with aspirin and ticagrelor are typically given for one year after index heart attack and then patients will continue to take aspirin lifelong. However, these patients are still having increased risk of suffering from another heart attack. Recently data showed that adding ticagrelor to aspirin in the long term can decrease the chance of recurrent heart attack but at the cost of increased risk of major bleeding. On the other hand, ticagrelor is a potent antiplatelet agent and has been showed to have additional benefit on blood vessels and platelets. The investigator hypothesize that monotherapy with ticagrelor may have further benefit over monotherapy with aspirin in the long term management in patients with history of heart attack. The investigator plan to perform a randomized study to compare the outcome in patients taking either ticagrelor or aspirin. The primary endpoint is measurement of endothelial function by flow mediated dilatation of brachial artery which is a surrogate marker of adverse cardiovascular outcome 3 months after treatment. The investigator would also investigate secondary endpoints of patients' blood level of adenosine activity, platelet function, endothelial progenitor cell count and biomarkers

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a disease with high mortality, morbidity and economic burden. Usually, it is caused by ischemic heart disease and atherosclerotic plaque rupture in the coronary arteries causing platelet activation, aggregation and thrombus formation. For decades, antiplatelet agents are the cornerstones of management of ACS and several clinical trials have confirmed greater clinical efficacy of dual antiplatelet therapy with clopidogrel and aspirin (ASA) versus ASA alone in patients with acute coronary syndromes (ACS) for up to a year of therapy. Ticagrelor (AZD6140) is a reversible, potent, oral adenosine diphosphate (ADP) P2Y12 receptor blocker which has stronger antiplatelet activity than clopidogrel. Data from PLATO, a Phase III pivotal efficacy and safety study of ticagrelor, have demonstrated superiority of ticagrelor 90 mg twice daily over clopidogrel 75 mg daily with a duration of up to 12 months in the prevention of fatal and non-fatal cardiovascular event in ACS patients on ASA.

In PLATO, ticagrelor was superior to clopidogrel in reducing the rate of the composite efficacy endpoint of CV death, MI, or stroke after ACS events. Furthermore, compared to clopidogrel, ticagrelor decreased the rate of death from any cause. PLATO-defined Major bleeding (primary safety endpoint) for ticagrelor did not differ significantly from that of clopidogrel but ticagrelor was associated with a higher rate of major bleeding not related to coronary-artery bypass grafting.

The favourable results lead to approval of use of ticagrelor as Class I indication in ACS patients for up to one year in addition to ASA in ACC/AHA and European guidelines. After one year of DAPT, patients typically remained on single antiplatelet agent with ASA monotherapy being the conventional treatment. However, these patients are still at heightened risk of recurrent atherothrombotic events. The recent PEGASUS TIMI 54 trial investigated the use of ticagrelor in addition to aspirin in stable patients with prior myocardial infarction one to three years ago. It demonstrated ticagrelor either 90mg BD or 60mg BD significantly reduced the risk of cardiovascular death, MI and stroke compared with placebo; ticagrelor 60mg BD. However, the use of ticagrelor is also associated with higher risks of major bleeding; ticagrelor 60mg BD, HR 2.32.

As the antithrombotic benefit of stronger antiplatelet effects of DAPT is offset by higher bleeding risk, it is reasonable to assume that a single potent antiplatelet agent such as ticagrelor may lead to better clinical outcome than ASA with less increase in bleeding risk when compared with DAPT. In addition to its antiplatelet effects, ticagrelor has been shown to improve endothelial function, increase plasma adenosine level, increase coronary blood flow, stabilize coronary plaques and reduce inflammation. These pleiotropic effects may lead to further clinical benefit of ticagrelor over other antiplatelet agents such as ASA and clopidogrel. Endothelial function as measured by flow mediated dilatation of brachial artery is a non-invasively measurable surrogate marker of adverse cardiovascular events. Adenosine is a purine nucleoside which has favourable effects on coronary vasodilatation, endothelial progenitor cell migration and ischemia-reperfusion injury while adenosine plasma activity can be measured by liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or above.
2. Documented history of presumed spontaneous ACS (excluding known peri-procedural or definite secondary MI [eg, due to profound hypotension, hypertensive emergency, tachycardia, or profound anemia]) with their most recent MI occurring 18 months or more prior to randomization
3. Patient currently prescribed and tolerating ASA
4. Females of child-bearing potential (ie, who are not chemically or surgically sterilized or who are not post-menopause) must have a negative urine pregnancy test at enrollment (to be confirmed by blood pregnancy test at the central lab.) Females of child-bearing potential must be willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator.
5. Written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Recurrent cardiovascular event (ACS, stroke and unplanned revascularization) after the index ACS
2. Planned use of ADP receptor blockers (eg, clopidogrel, ticlopidine, prasugrel), dipyridamole, or cilostazol
3. Planned coronary, cerebrovascular, or peripheral arterial revascularization
4. Concomitant oral or intravenous therapy with strong cytochrome P450 3A (CYP3A) inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers which cannot be stopped for the course of the study - Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir, over 1 litre daily of grapefruit juice - Substrates with narrow therapeutic index: cyclosporine, quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily
5. Concomitant use of vasoactive drugs or vasoactive drugs cannot be stopped.
6. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin (at venous thrombosis treatment not prophylaxis doses)
7. Patients with known bleeding diathesis or coagulation disorder
8. Patients with:

   * Concomitant active pathological bleeding,
   * A history of intracranial bleed at any time,
   * A central nervous system tumour or intracranial vascular abnormality (eg, aneurysm, arteriovenous malformation) at any time,
   * Intracranial or spinal cord surgery within 5 years, or
   * A gastrointestinal (GI) bleed within the past 6 months, or major surgery within 30 days
9. History of ischemic stroke at any time
10. Patients considered to be at risk of bradycardic events ([eg, known sick sinus syndrome or second or third degree atrioventricular (AV) block]) unless already treated with a permanent pacemaker
11. Coronary-artery bypass grafting in the past 5 years, unless the patient has experienced a spontaneous MI subsequent to the bypass surgery.
12. Known severe liver disease (eg, ascites or signs of coagulopathy)
13. Renal failure requiring dialysis or anticipated need for dialysis during the course of the study
14. Hypersensitivity to ticagrelor or any excipients
15. Pregnancy or lactation
16. Life expectancy < 1 year
17. Any condition which in the opinion of the Investigator would make it unsafe or unsuitable for the patient to participate in this study (eg, active malignancy other than squamous cell or basal cell skin cancer)
18. Concern for inability of the patient to comply with study procedures and/or follow up (eg, alcohol or drug abuse)
19. Participation in previous study with ticagrelor if treated with ticagrelor. Previous randomization in the present study
20. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
21. Participation in another clinical study with an investigational product during the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 3 months
  the flow mediated dilatation of brachial artery at baseline and 3 months after randomization. Demonstrate brachial diameters, the measurement will be presented in absolute FMD millimeter (FMDmm). The report value should be present in FMD percentage (FMD%) as the mean of baseline measurement minus the mean of 3 months measurement then divided by the 3 months measurement.

SECONDARY OUTCOMES:
Plasma adenosine level Platelet function parameters Endothelial progenitor cell count Biomarkers such as highly sensitive troponin | 3 months
  collect the blood sample to test the Plasma adenosine level Platelet function parameters Endothelial progenitor cell count Biomarkers such as highly sensitive troponin at baseline and 3 months after randomization. The unit of the test should be nmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. HF Tse, Hong Kong, China

REFERENCES:
- [Result] Chen ZM, Jiang LX, Chen YP, Xie JX, Pan HC, Peto R, Collins R, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Addition of clopidogrel to aspirin in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1607-21. doi: 10.1016/S0140-6736(05)67660-X. PMID 16271642
- [Result] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Bonaca MP, Bhatt DL, Cohen M, Steg PG, Storey RF, Jensen EC, Magnani G, Bansilal S, Fish MP, Im K, Bengtsson O, Oude Ophuis T, Budaj A, Theroux P, Ruda M, Hamm C, Goto S, Spinar J, Nicolau JC, Kiss RG, Murphy SA, Wiviott SD, Held P, Braunwald E, Sabatine MS; PEGASUS-TIMI 54 Steering Committee and Investigators. Long-term use of ticagrelor in patients with prior myocardial infarction. N Engl J Med. 2015 May 7;372(19):1791-800. doi: 10.1056/NEJMoa1500857. Epub 2015 Mar 14. PMID 25773268
- [Result] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members; Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):2354-94. doi: 10.1161/CIR.0000000000000133. Epub 2014 Sep 23. No abstract available. PMID 25249586
- [Result] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Result] Cattaneo M, Schulz R, Nylander S. Adenosine-mediated effects of ticagrelor: evidence and potential clinical relevance. J Am Coll Cardiol. 2014 Jun 17;63(23):2503-2509. doi: 10.1016/j.jacc.2014.03.031. Epub 2014 Apr 23. PMID 24768873
- [Result] Inaba Y, Chen JA, Bergmann SR. Prediction of future cardiovascular outcomes by flow-mediated vasodilatation of brachial artery: a meta-analysis. Int J Cardiovasc Imaging. 2010 Aug;26(6):631-40. doi: 10.1007/s10554-010-9616-1. Epub 2010 Mar 26. PMID 20339920
- [Result] Ras RT, Streppel MT, Draijer R, Zock PL. Flow-mediated dilation and cardiovascular risk prediction: a systematic review with meta-analysis. Int J Cardiol. 2013 Sep 20;168(1):344-51. doi: 10.1016/j.ijcard.2012.09.047. Epub 2012 Oct 4. PMID 23041097
- [Result] Bonello L, Laine M, Kipson N, Mancini J, Helal O, Fromonot J, Gariboldi V, Condo J, Thuny F, Frere C, Camoin-Jau L, Paganelli F, Dignat-George F, Guieu R. Ticagrelor increases adenosine plasma concentration in patients with an acute coronary syndrome. J Am Coll Cardiol. 2014 Mar 11;63(9):872-7. doi: 10.1016/j.jacc.2013.09.067. Epub 2013 Nov 27. PMID 24291273
- [Result] Bhatt DL, Steg PG, Ohman EM, Hirsch AT, Ikeda Y, Mas JL, Goto S, Liau CS, Richard AJ, Rother J, Wilson PW; REACH Registry Investigators. International prevalence, recognition, and treatment of cardiovascular risk factors in outpatients with atherothrombosis. JAMA. 2006 Jan 11;295(2):180-9. doi: 10.1001/jama.295.2.180. PMID 16403930
- [Derived] Tam CF, Chan YH, Wong YK, Li Z, Zhu X, Su KJ, Ganguly A, Hwa K, Ling XB, Tse HF. Multi-Omics Signatures Link to Ticagrelor Effects on Vascular Function in Patients With Acute Coronary Syndrome. Arterioscler Thromb Vasc Biol. 2022 Jun;42(6):789-798. doi: 10.1161/ATVBAHA.121.317513. Epub 2022 Apr 7. PMID 35387483